CLINICAL TRIAL: NCT02168790
Title: Interventional Study to Investigate the Safety of a Combination of Amniotic Membrane and a Holder Device (AmnioClip) in the Therapy of Ocular Surface Disorders (Sutureless Amniotic Membrane Transplantation)
Brief Title: Safety Study of a Sutureless Amniotic Membran Transplantation to Treat Ocular Surface Disorders (Expanded Access)
Acronym: AmnioClip
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Klinikum Chemnitz gGmbH (Other)
Collaborators: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Katrin Engelmann, Principal Investigator, Klinikum Chemnitz gGmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKC002AR01
Record Dates: First submitted 2014-06-12; First posted 2014-06-20 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Corneal Ulcers; Corneal Melting
Keywords: amniotic membrane holder, aminiotic membrane transplantation
MeSH Terms: conditions — Corneal Ulcer | interventions — Biological Dressings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amniotic membrane ring (Experimental): Application of amniotic membrane device for 6-7 days.
  Interventions: Device: Amniotic membrane ring

INTERVENTIONS:
Device: Amniotic membrane ring — The amniotic membrane ring system (AmnioClip) is device for sutureless application of amniotic membrane to oculare surfaces. Amniotic membrane is mounted between the two rings with a specially designed, accessory mounting device.
  Other Names: Amniotic membrane

SUMMARY:
The investigators aimed at developing a technique to apply amniotic membrane to a diseased ocular surface without surgical intervention (sutureless amniotic membrane transplantation). This system needs to be concordant with laws and guidelines for the use of medical and pharmaceutical products.

DETAILED DESCRIPTION:
A ring system (AmnioClip) was developed for mounting an amniotic membrane (AM) that can be applied like a large contact lens. AM is mounted between the two rings with a special designed, accessory mounting device. The safety of the ring system AmnioClip was tested in an interventional including 7 patients with ocular surface disorders and need for AM transplantation (1, 2, 3). About similar systems was reported (3, 4).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ocular surface disorders and indication for amniotic membrane transplantation
* Willingness to provide signed Informed Consent Form
* For sexually active women of childbearing potential, use of an appropriate form of contraception (or abstinence) for the duration of the study
* Ability and willingness to return for all scheduled visits and assessments

Exclusion Criteria:

* An eye that, in the investigator's opinion, would not benefit from amniotic membrane transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Slit lamp investigation of the inflammation status of the conjunctiva | Participants will be followed for the duration of hospital stay, an expanded average of 3 month
  The ring of the AmnioClip touches the conjunctiva of the ocular surface. To prove side effects through the medical device the conjunctiva is controlled at every visit with microscopy using a slit lamp.

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Kotomin, Study Chair — Klinikum Chemnitz gGmbH
Locations (1):
- Klinikum Chemnitz gGmbH, Chemnitz, Saxony, Germany

REFERENCES:
- [Background] 1. Liu J, Sheha H, Fu Y et al. (2010) Update of amniotic membrane transplantation. Expert Review Ophthalmol 5:645-661 2. Dua HS, Azuara-Blanco A (1999) Amniotic membrane transplantation, Br J Ophthalmol 83:748-752 3. Daniel Meller, Mikk Pauklin, Henning Thomasen et al. (2011) Amniotic Membrane Transplantation in the Human Eye. Dtsch Arztebl Int 108: 243-8 4. Pachigolla G, Prasher P, Di Pasauale MA, Mc Culley JP, Mc Henry JG, Mootha VV, Evaluation of the role of ProKera in the mamagment of ocular surface and orbital disorders, Eye Contact Lens 2009, 35:172-175 5. Uhlig CE and Busse H, Development and evaluation of a device for sutureless and repeated application of amniotic memnbrane overlays. Cornea 29:331-5
- [Derived] Kotomin I, Valtink M, Hofmann K, Frenzel A, Morawietz H, Werner C, Funk RH, Engelmann K. Sutureless fixation of amniotic membrane for therapy of ocular surface disorders. PLoS One. 2015 May 8;10(5):e0125035. doi: 10.1371/journal.pone.0125035. eCollection 2015. PMID 25955359